CLINICAL TRIAL: NCT02025556
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Study Comparing the Efficacy and Safety of Two Doses of Subcutaneous LBR-101 With Placebo for the Preventive Treatment of High Frequency Episodic Migraine
Brief Title: A Multicenter Assessment of LBR-101 in High Frequency Episodic Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: NCGS, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LBR-101-022
Record Dates: First submitted 2013-12-20; First posted 2014-01-01 (Estimated); Results first posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Episodic Migraine Headache
Keywords: High Frequency Episodic Migraine Headache; Episodic Migraine Headache; Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — fremanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LBR-101 High Dose (Experimental): Subcutaneous High Dose LBR-101 Administered Monthly x 3
  Interventions: Drug: LBR-101 High Dose
- LBR-101 Low Dose (Experimental): Subcutaneous Low Dose LBR-101 Administered Monthly x 3
  Interventions: Drug: LBR-101 Low Dose
- Placebo (Placebo Comparator): Subcutaneous Placebo Administered Monthly x 3
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LBR-101 High Dose — Subcutaneously Administered High Dose LBR-101 Monthly x 3
  Other Names: Fremanezumab
  Arms: LBR-101 High Dose
Drug: LBR-101 Low Dose — Subcutaneously Administered Low Dose LBR-101 Monthly x 3
  Other Names: Fremanezumab
  Arms: LBR-101 Low Dose
Drug: Placebo — Subcutaneously Administered Placebo (Vehicle) Monthly x 3
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether monthly subcutaneous administration of LBR-101 (fremanezumab) is safe and provides migraine prevention in subjects with high frequency episodic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 65 years of age.
* A signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study including any known and potential risks and available alternative treatments.
* Subjects fulfilling criteria for episodic migraine as per the Second Edition of The International Headache Society (Olesen and Steiner 2004), who experience migraine at high frequency as follows:

  i. History of headaches on more than 8 days per month for at least 3 months prior to screening

ii. Verification of headache frequency through prospectively collected baseline information during the 28-day run-in phase demonstrating headaches (of any type) on at least 8 days with at total of 8 to 14 days* fulfilling criteria for migraine.

*Operational definition for migraine and probable migraine days are presented in the statistical section of this protocol.

* Body Mass Index (BMI) of 17.5 to 37.5 kg/m2, and a total body weight between 50 kg and 120 kg, inclusive.
* Demonstrated compliance with the electronic headache diary during the run-in period by entry of headache data on a minimum of 22/28 days (80% compliance).

Exclusion Criteria:

* Subject has received onabotulinum toxin A for migraine or for any medical or cosmetic reasons requiring injections in the head, face, or neck during the six months prior to screening.
* Subject uses medications containing opioids (including codeine) or barbiturates (including Fiorinal®, Fioricet®, or any other combination containing butalbital) on more than 4 days per month for the treatment of migraine or for any other reason.
* Failed > 2 medication categories or > 3 preventive medications (within two medication categories) due to lack of efficacy for prophylactic treatment of episodic or chronic migraine after an adequate therapeutic trial
* Treatment with an investigational drug or device within 30 days of study entry or any prior exposure to a monoclonal antibody targeting the CGRP pathway.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2015-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Pharmaceuticals USA
Locations (63):
- United States (63):
  - Teva Investigational Site 145, Gilbert, Arizona
  - Teva Investigational Site 130, Phoenix, Arizona
  - Teva Investigational Site 117, Scottsdale, Arizona
  - Teva Investigational Site 158, Little Rock, Arkansas
  - Teva Investigational Site 161, Anaheim, California
  - Teva Investigational Site 116, Fullerton, California
  - Teva Investigational Site 119, Long Beach, California
  - Teva Investigational Site 146, Oceanside, California
  - Teva Investigational Site 113, San Francisco, California
  - Teva Investigational Site 108, Stanford, California
  - Teva Investigational Site 112, Walnut Creek, California
  - Teva Investigational Site 132, Boulder, Colorado
  - Teva Investigational Site 162, Stamford, Connecticut
  - Teva Investigational Site 143, DeLand, Florida
  - Teva Investigational Site 137, Hialeah, Florida
  - Teva Investigational Site 159, Hollywood, Florida
  - Teva Investigational Site 101, Jacksonville, Florida
  - Teva Investigational Site 166, Jacksonville, Florida
  - Teva Investigational Site 129, Maitland, Florida
  - Teva Investigational Site 167, Orlando, Florida
  - Teva Investigational Site 139, Ormond Beach, Florida
  - Teva Investigational Site 140, Port Orange, Florida
  - Teva Investigational Site 160, South Miami, Florida
  - Teva Investigational Site 149, Atlanta, Georgia
  - Teva Investigational Site 164, Decatur, Georgia
  - Teva Investigational Site 134, Douglasville, Georgia
  - Teva Investigational Site 125, Evansville, Indiana
  - Teva Investigational Site 133, Lenexa, Kansas
  - Teva Investigational Site 135, Brockton, Massachusetts
  - Teva Investigational Site 124, New Bedford, Massachusetts
  - Teva Investigational Site 151, Springfield, Massachusetts
  - Teva Investigational Site 109, Watertown, Massachusetts
  - Teva Investigational Site 115, Worcester, Massachusetts
  - Teva Investigational Site 110, Ann Arbor, Michigan
  - Teva Investigational Site 114, Kalamazoo, Michigan
  - Teva Investigational Site 150, Golden Valley, Minnesota
  - Teva Investigational Site 152, Kansas City, Missouri
  - Teva Investigational Site 107, Springfield, Missouri
  - Teva Investigational Site 104, St Louis, Missouri
  - Teva Investigational Site 148, Reno, Nevada
  - Teva Investigational Site 105, The Bronx, New York
  - Teva Investigational Site 131, Greensboro, North Carolina
  - Teva Investigational Site 118, Raleigh, North Carolina
  - Teva Investigational Site 165, Raleigh, North Carolina
  - Teva Investigational Site 168, Winston-Salem, North Carolina
  - Teva Investigational Site 122, Canton, Ohio
  - Teva Investigational Site 141, Cincinnati, Ohio
  - Teva Investigational Site 142, Cincinnati, Ohio
  - Teva Investigational Site 155, Cleveland, Ohio
  - Teva Investigational Site 102, Columbus, Ohio
  - Teva Investigational Site 127, Oklahoma City, Oklahoma
  - Teva Investigational Site 111, Philadelphia, Pennsylvania
  - Teva Investigational Site 120, Goose Creek, South Carolina
  - Teva Investigational Site 153, Bristol, Tennessee
  - Teva Investigational Site 126, Memphis, Tennessee
  - Teva Investigational Site 154, Nashville, Tennessee
  - Teva Investigational Site 128, Arlington, Texas
  - Teva Investigational Site 121, Austin, Texas
  - Teva Investigational Site 136, Austin, Texas
  - Teva Investigational Site 156, Mansfield, Texas
  - Teva Investigational Site 157, Salt Lake City, Utah
  - Teva Investigational Site 123, Charlottesville, Virginia
  - Teva Investigational Site 144, Roanoke, Virginia

REFERENCES:
- [Derived] Silberstein SD, Rapoport AM, Loupe PS, Aycardi E, McDonald M, Yang R, Bigal ME. The Effect of Beginning Treatment With Fremanezumab on Headache and Associated Symptoms in the Randomized Phase 2 Study of High Frequency Episodic Migraine: Post-Hoc Analyses on the First 3 Weeks of Treatment. Headache. 2019 Mar;59(3):383-393. doi: 10.1111/head.13446. Epub 2018 Nov 18. PMID 30450545
- [Derived] VanderPluym J, Dodick DW, Lipton RB, Ma Y, Loupe PS, Bigal ME. Fremanezumab for preventive treatment of migraine: Functional status on headache-free days. Neurology. 2018 Sep 18;91(12):e1152-e1165. doi: 10.1212/01.wnl.0000544321.19316.40. Epub 2018 Aug 17. PMID 30120138
- [Derived] Halker Singh RB, Aycardi E, Bigal ME, Loupe PS, McDonald M, Dodick DW. Sustained reductions in migraine days, moderate-to-severe headache days and days with acute medication use for HFEM and CM patients taking fremanezumab: Post-hoc analyses from phase 2 trials. Cephalalgia. 2019 Jan;39(1):52-60. doi: 10.1177/0333102418772585. Epub 2018 May 3. PMID 29722276
- [Derived] Cohen JM, Dodick DW, Yang R, Newman LC, Li T, Aycardi E, Bigal ME. Fremanezumab as Add-On Treatment for Patients Treated With Other Migraine Preventive Medicines. Headache. 2017 Oct;57(9):1375-1384. doi: 10.1111/head.13156. Epub 2017 Sep 1. PMID 28862758
- [Derived] Bigal ME, Dodick DW, Rapoport AM, Silberstein SD, Ma Y, Yang R, Loupe PS, Burstein R, Newman LC, Lipton RB. Safety, tolerability, and efficacy of TEV-48125 for preventive treatment of high-frequency episodic migraine: a multicentre, randomised, double-blind, placebo-controlled, phase 2b study. Lancet Neurol. 2015 Nov;14(11):1081-90. doi: 10.1016/S1474-4422(15)00249-5. Epub 2015 Sep 30. PMID 26432182

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 297 participants with episodic migraine were enrolled in the study.
Pre-assignment Details: Participants were assigned to receive either subcutaneous administration of 675 mg of fremanezumab (LBR-101) for three months, subcutaneous administration of 225 mg of fremanezumab (LBR-101) for three months, or subcutaneous administration of placebo for three months.
Groups:
- Placebo: Participants received subcutaneous placebo injections at one visit per month for three months (Day
  1/week 0, Day 29/week 4, and Day 57/week 8).
- Low Dose: Participants received 225 mg fremanezumab subcutaneously on Day 1/week 0, Day 29/week 4, and on Day 57/week 8.
- High Dose: Participants received 675 mg fremanezumab subcutaneously on Day 1/week 0, Day 29/week 4, and on Day 57/week 8.
Period: Overall Study
Arm/Group | Placebo | Low Dose | High Dose
Started (All randomized participants) | 104 | 96 | 97
Safety Analysis Set (All randomized participants who received at least one dose of study drug) | 104 | 96 | 96
Intent-to-treat (ITT) Set (Received at least one dose of study drug and obtained at least one efficacy measurement) | 104 | 95 | 96
Completed | 98 | 83 | 88
Not Completed | 6 | 13 | 9
Not completed — Adverse Event | 0 | 4 | 2
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 6
Not completed — Lost to Follow-up | 2 | 4 | 0
Not completed — Reason not reported | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose | High Dose | Total
Number analyzed (Participants) | 104 | 96 | 97 | 297
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.0 (11.62) | 40.8 (12.43) | 40.7 (12.56) | 41.2 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 87 | 82 | 261
  Male | 12 | 9 | 15 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 16 | 17 | 44
  Not Hispanic or Latino | 92 | 80 | 79 | 251
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 19 | 18 | 50
  White | 85 | 74 | 74 | 233
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 4 | 10
Years of migraine [Mean (Standard Deviation); unit: Years] | 21.2 (14.1) | 18.9 (12.92) | 16.9 (12.25) | 19.0 (13.21)
Preventive medication use [Count of Participants; unit: Participants] — Participants reported preventive migraine medication use at the time of randomization
  Participants
    Yes | 28 | 32 | 26 | 86
    No | 76 | 64 | 71 | 211

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Monthly Migraine Days During the 28-day Post Treatment Period Ending With Week 12
Description: A migraine day was endorsed when at least 1 of the following situations occurred: 1) A calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache endorsing criteria for migraine, or 2) a calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache endorsing criteria for probable migraine, a migraine subtype where only one migraine criterion is missing, or 3) the participant used acute migraine medication (triptans and ergot compounds) to treat a headache of any duration, or 4) any of the above days preceded or followed by a day with a headache of any duration. This calculation was defined as the change from baseline in the number of headache days during the 28-day post treatment period ending at week 12. Headache severity was rated daily by the participant as either no pain, mild, moderate, or severe.
Time Frame: Baseline to week 12
Population: Intent-to-treat (ITT) population includes all randomized participants that received at least one dose and obtained at least one endpoint measurement.
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo | Low Dose | High Dose
Number analyzed (Participants) | 104 | 95 | 96
Days | -3.46 (0.53) | -6.27 (0.55) | -6.09 (0.53)
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority; p < .0001, Mixed Models Analysis — The threshold for statistical significance was p = .05; Mean Difference (Final Values) = -2.81, 95% CI 2-sided [-4.07 to -1.55], Standard Error of Mean 0.64
Statistical Analysis 2: Comparison: Placebo vs High Dose; Test type: Superiority; p < .0001, Mixed Models Analysis — The threshold for statistical significance was p = .05; Mean Difference (Final Values) = -2.64, 95% CI 2-sided [-3.9 to -1.38], Standard Error of Mean 0.64

2. Primary Outcome: Number of Participants With at Least One Adverse Event
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Relationship of AE to treatment was determined by the Investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent the previously listed serious outcomes. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline to week 12
Population: Safety analysis set included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Placebo | Low Dose | High Dose
Number analyzed (Participants) | 104 | 96 | 96
Participants | 58 | 44 | 57

3. Primary Outcome: Number of Participants Reporting Mild, Moderate, and Severe Adverse Events (AEs)
Description: Adverse events were rated based on the investigator's clinical judgment. Mild: awareness of a sign or symptom that was easily tolerated Moderate: sign or symptom intense enough to interfere with usual activity Severe: interfered significantly with ability to do work or usual activity
Time Frame: Up to week 12
Population: Per planned analysis participants analyzed included all randomized participants who received at least one dose of study drug and reported at least one adverse event.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low Dose | High Dose
Number analyzed (Participants) | 58 | 44 | 57
Participants
  Mild | 29 | 20 | 31
  Moderate | 27 | 20 | 26
  Severe | 1 | 4 | 0
  Unknown severity | 1 | 0 | 0

4. Secondary Outcome: Change From Baseline in Number of Days With Headache of Any Severity
Description: A headache day was defined as when at least 1 of the following situations occurred: A calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours of a headache of any severity or the participant used acute migraine medication (triptans and ergot compounds) to treat a headache. This calculation was defined as the change from baseline in the number of headache days during the 28-day post treatment period ending at week 12. Headache severity was rated daily by the participant as either no pain, mild, moderate, or severe.
Time Frame: Baseline to week 12
Population: Intent-to-treat (ITT) population includes all randomized participants who received at least one dose of study medication and obtained at least one endpoint measurement.
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo | Low Dose | High Dose
Number analyzed (Participants) | 104 | 95 | 96
Days | -3.52 (0.53) | -6.14 (0.56) | -6.10 (0.54)

ADVERSE EVENTS:
Time Frame: Baseline to week 12
Arm/Group | Placebo | Low Dose | High Dose
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/96 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/104 | 2/96 | 2/96
Other Adverse Events (participants affected / at risk) | 9/104 | 9/96 | 11/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=104) | Low Dose (N=96) | High Dose (N=96)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=104) | Low Dose (N=96) | High Dose (N=96)
Injection site pain (General disorders) | 6 (10) | 9 (13) | 4 (4)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 5 (5)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.